CLINICAL TRIAL: NCT00327899
Title: Home Inotropic Therapy in Children
Status: Terminated | Type: Observational
Why Stopped: Per PI instruction.
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 06-129
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2007-11

CONDITIONS: Congenital Disorders
Keywords: pediatric; congestive heart failure; inotropes
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Heart Failure

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Inotropic therapy is a well-established practice for children with advanced congestive heart failure (CHF). Inotropes are intravenous medications to help the heart pump stronger and prolong life while awaiting heart transplantation. Traditionally children have been maintained on inotropic therapy in the hospital under close, monitored supervision. The United Network for Organ Sharing (UNOS), which governs organ distribution, has now changed listing criteria allowing patients awaiting heart transplantation to be discharged to home, yet maintaining a higher status on the waiting list. In adults, home inotropic therapy has been shown to be a safe and cost-effective bridge to transplantation. To date, there are no data on the use of home inotropic therapy in children.

Hypothesis:

We request to do a retrospective chart review of patients receiving this therapy to determine safety and efficacy of continuous ambulatory home inotropic therapy in children.

DETAILED DESCRIPTION:
Hypothesis:

We request to do a retrospective chart review of patients receiving this therapy to determine safety and efficacy of continuous ambulatory home inotropic therapy in children.

Methods:

Data will be obtained from CHOA and Coram Home Healthcare, Inc over a two year period, January 1, 2004 through December 31, 2005. Data will be collected on approximately 35 children aged 0-18 years receiving therapy. The length of therapy, type of therapy, therapy-related complications, number of readmissions, deaths at home and catheter-related infections data will be collected.

Inclusion Criteria:

Receiving inotropic support at home Choa patients with Coram Healthcare only

ELIGIBILITY:
Inclusion Criteria:

* Receiving inotropic support at home
* Choa patients with Coram Healthcare only
* medical charts between 2.2.2004 and 12.31.2005

Exclusion Criteria:

* those who do not meet inclusion criteria

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Choa patients' medical charts between 2.2.04 and 12.31.05 with Coram Healthcare only. These patients would have received inotropic support at home.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2006-03; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandria Berg, MSN, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States